CLINICAL TRIAL: NCT04060069
Title: Influence of Pneumoperitoneum and Trendelenburg Position on Fluid Responsiveness Predicted by Pulse Pressure Variation and Stroke Volume Variation During Anaesthesia for Laparoscopic Gynaecological Surgery
Brief Title: Pneumoperitoneum and Trendelenburg Position on Fluid Responsiveness
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Tulay Sahin, Clinical Professor, Kocaeli University
Other Study IDs: KOU GOKAEK 2016/272
Record Dates: First submitted 2019-08-09; First posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Fluid Responsiveness
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Before pneumoperitoneum: Fluid administration
  Interventions: Other: Ringer Lactate

INTERVENTIONS:
Other: Ringer Lactate — Fluids

SUMMARY:
The increased intraabdominal pressure and intrathoracic pressure due to pneumoperitoneum negatively affect the cardiovascular system, relatively dynamic parameters may vary due to intraoperative fluid therapy.

DETAILED DESCRIPTION:
After the general anaesthesia induction and intubation, dynamic parameters such as SVV and PPV were monitored by pulse contour analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old patients
* Will undergo elective laparoscopic gynecological surgery
* ASA I-II

Exclusion Criteria:

* Obese patients (body mass index> 30 kg.m2)
* Patients who had arrhythmia
* Patients who had cardiac insufficiency.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 45 patients over the age of 18 who would undergo elective laparoscopic gynecological surgery and had the ASA (American Society of Anesthesiologists) risk classification I-II were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
to evaluate how stroke volume variation (%) affected during the Trendelenburg position and pneumoperitoneum | up to 10 months
  to evaluate reliability of stroke volume variation in evaluating the response to fluid administration
to evaluate how pulse pressure variation (%) affected during the Trendelenburg position and pneumoperitoneum | up to 10 months
  to evaluate reliability of pulse pressure variation in evaluating the response to fluid administration